CLINICAL TRIAL: NCT03185065
Title: Treatment of Fatigue With Methylphenidate, Modafinil and Amantadine in Multiple Sclerosis
Acronym: TRIUMPHANT-MS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00119702
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Fatigue in Multiple Sclerosis
MeSH Terms: interventions — Amantadine; Modafinil; Methylphenidate

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled, crossover, 4-sequence, 4-period, double-blind, multicenter trial of 3 commonly used medications for treatment of Multiple Sclerosis related fatigue versus placebo in fatigued subjects with MS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (Experimental): amantadine, placebo, modafinil, methylphenidate
  Interventions: Drug: Amantadine; Drug: Modafinil; Drug: Methylphenidate; Drug: Placebos
- Arm B (Experimental): placebo, methylphenidate, amantadine, modafinil
  Interventions: Drug: Amantadine; Drug: Modafinil; Drug: Methylphenidate; Drug: Placebos
- Arm C (Experimental): modafinil, amantadine, methylphenidate, placebo
  Interventions: Drug: Amantadine; Drug: Modafinil; Drug: Methylphenidate; Drug: Placebos
- Arm D (Experimental): methylphenidate, modafinil, placebo and amantadine
  Interventions: Drug: Amantadine; Drug: Modafinil; Drug: Methylphenidate; Drug: Placebos

INTERVENTIONS:
Drug: Amantadine — 100 mg of amantadine increased to 200 mg of amantadine, if tolerated
Drug: Modafinil — 100 mg of modafinil increased to 200 mg of modafinil, if tolerated
Drug: Methylphenidate — 5 mg of methylphenidate uptitrated to max of 20 mg of methylphenidate, if tolerated
Drug: Placebos — 1 placebo capsule increased to max of 2 capsules twice daily

SUMMARY:
Randomized, placebo-controlled, crossover, 4-sequence, 4-period, double-blind (participants and investigators), multicenter trial of 3 commonly used medications for treatment of MS-related fatigue (amantadine, modafinil, methylphenidate) versus placebo in fatigued subjects with MS defined by McDonald Criteria.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, crossover, 4-sequence, 4-period, double-blind (participants and investigators), multicenter trial of 3 commonly used medications for treatment of MS-related fatigue (amantadine, modafinil, methylphenidate) versus placebo in fatigued subjects with MS defined by McDonald Criteria.

Using a balanced Latin-square crossover design, subjects will be allocated, in a double-blind, randomized fashion, to one of the four treatment sequences (Figure 1): 1) amantadine, placebo, modafinil, methylphenidate; 2) placebo, methylphenidate, amantadine, modafinil; 3) modafinil, amantadine, methylphenidate, placebo; and 4) methylphenidate, modafinil, placebo and amantadine. Each medication will be titrated over four weeks to the participants' highest tolerated dose or the pre-defined highest dose. The dosing and titration schedule of the study medications are depicted in Figure 2. Each treatment period will be 6 weeks and there will be a 2-week washout period between each treatment period. At the beginning of the trial, a biostatistician at University of California, San Francisco (UCSF) will prepare a concealed allocation schedule, randomly assigning the four sequences, in blocks of 4, to a consecutive series of numbers and at the time of enrollment, each participant will be assigned the next consecutive number (and hence the sequence of study medications).

The primary endpoint of the study will be fatigue severity as measured by the MFIS score, between 26th and 35th day of each treatment period (while the patient is taking the maximal tolerated or target dose). The MFIS is a validated patient-reported outcome. The questionnaire will be administered remotely (through internet, phone or mailed forms) and the participants can answer the questions in few minutes while at home or at their work place. The questionnaire has been validated in English and Spanish.

ELIGIBILITY:
Inclusion criteria:

* Age 18 years and older.
* Females of childbearing age must have a negative urine pregnancy test at baseline and use an effective method of contraception during the study.
* Diagnosis of MS (according to the 2010 McDonald criteria).
* Expanded Disability Status Scale (EDSS) score at the time of screening 0.0-7.0.
* Fatigue reportedly present and screening Modified Fatigue Impact Scale (MFIS) score more than 33.
* At least a two-week washout for any fatigue-related drug, including study medications.

Exclusion criteria:

* Neurodegenerative disorders other than relapsing or progressive MS.
* Breastfeeding or pregnant.
* History of coronary artery disease or congestive heart failure.
* Uncontrolled hypertension at screening (history of high blood pressure and screening systolic blood pressure >160 or diastolic blood pressure>100).
* Glomerular Filtration Rate (GFR) (glomerular filtration rate) < 50.
* Abnormal liver function at screening (AST or Alanine Aminotransferase (ALT) more than twice the upper limit of normal).
* Terminal medical conditions.
* Currently treated for active malignancy.
* Planned surgery or move within 8 months of screening.
* Alcohol or substance abuse in the past year (except marijuana or other cannabinoids).
* A history of intolerance or allergic or anaphylactic reaction to amantadine, modafinil, methylphenidate or any component of the preparation.
* Clinically unstable medical or psychiatric disorders that require acute treatment as determined by the PI.
* Concurrent use of monoamine oxidase inhibitors-B.
* Hypersensitivity/idiosyncrasy to sympathomimetic amines
* Inability to communicate or answer the questionnaires in English or Spanish.
* Severe untreated anemia (blood hemoglobin <9gr/dl)
* History of untreated hypothyroidism
* History of untreated sleep apnea
* History of long QT syndrome, atrial fibrillation or tachyarrhythmias (other than sinus tachycardia)
* History of ischemic or hemorrhagic stroke
* History of glaucoma
* History of Tourette syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bardia Nourbakhsh, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nourbakhsh B, Revirajan N, Morris B, Cordano C, Creasman J, Manguinao M, Krysko K, Rutatangwa A, Auvray C, Aljarallah S, Jin C, Mowry E, McCulloch C, Waubant E. Safety and efficacy of amantadine, modafinil, and methylphenidate for fatigue in multiple sclerosis: a randomised, placebo-controlled, crossover, double-blind trial. Lancet Neurol. 2021 Jan;20(1):38-48. doi: 10.1016/S1474-4422(20)30354-9. Epub 2020 Nov 23. PMID 33242419
- [Derived] Nourbakhsh B, Revirajan N, Waubant E. Treatment of fatigue with methylphenidate, modafinil and amantadine in multiple sclerosis (TRIUMPHANT-MS): Study design for a pragmatic, randomized, double-blind, crossover clinical trial. Contemp Clin Trials. 2018 Jan;64:67-76. doi: 10.1016/j.cct.2017.11.005. Epub 2017 Nov 4. PMID 29113955

RESULTS

PARTICIPANT FLOW:
Period: Period 1 (6 Weeks)
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 35 | 34 | 35 | 37
Completed | 32 | 33 | 32 | 36
Not Completed | 3 | 1 | 3 | 1
Period: Washout (2 Weeks)
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 32 | 33 | 32 | 36
Completed | 32 | 31 | 32 | 35
Not Completed | 0 | 2 | 0 | 1
Period: Period 2 (6 Weeks)
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 32 | 31 | 32 | 35
Completed | 32 | 31 | 32 | 34
Not Completed | 0 | 0 | 0 | 1
Period: Washout (2 Weeks)
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 32 | 31 | 32 | 34
Completed | 31 | 29 | 31 | 32
Not Completed | 1 | 2 | 1 | 2
Period: Period 3 (6 Weeks)
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 31 | 29 | 31 | 32
Completed | 31 | 29 | 29 | 32
Not Completed | 0 | 0 | 2 | 0
Period: Washout (2 Weeks)
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 31 | 29 | 29 | 32
Completed | 31 | 28 | 27 | 32
Not Completed | 0 | 1 | 2 | 0
Period: Period 4 (6 Weeks)
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 31 | 28 | 27 | 32
Completed | 31 | 27 | 26 | 31
Not Completed | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Total
Number analyzed (Participants) | 35 | 34 | 35 | 37 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (9.9) | 46.9 (12.4) | 46.1 (10.3) | 45.8 (10.2) | 46.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 27 | 29 | 109
  Male | 8 | 8 | 8 | 8 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 5 | 4 | 19
  White | 27 | 25 | 26 | 29 | 107
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 4 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Modified Fatigue Impact Scale (MFIS) Score
Description: MFIS score during the fifth week of treatment period. The total score of the MFIS ranges from 0 to 84. Higher scores denote more severe fatigue.
Time Frame: Week 5 of each treatment period
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Placebo: 1 placebo capsule increased to max of 2 capsules twice daily
Arm/Group | Placebo | Amantadine | Modafinil | Methylphenidate
Number analyzed (Participants) | 123 | 124 | 124 | 127
score on a scale | 40.6 [38.2 to 43.1] | 41.3 [38.8 to 43.7] | 39.0 [36.6 to 41.4] | 38.6 [36.2 to 41.0]

2. Secondary Outcome: Quality of Life in Neurological Disorders (Neuro-QoL) Item Bank - Fatigue Score
Description: Neuro-QoL Item Bank - Fatigue T score during the fifth week of treatment period. T-score distributions rescale raw scores into standardized scores with a mean of 50 and a standard deviation (SD) of 10. Higher T-scores denote more severe fatigue.
Time Frame: Week 5 of each treatment period
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Amantadine | Modafinil | Methylphenidate
Number analyzed (Participants) | 123 | 124 | 124 | 127
score on a scale | 53.1 [51.9 to 54.3] | 53.0 [51.7 to 54.2] | 52.5 [51.3 to 53.8] | 52.0 [50.8 to 53.2]

3. Secondary Outcome: Epworth Sleepiness Scale (ESS) Score
Description: ESS score during the fifth week of treatment period. The ESS score can range from 0 to 24. The higher the score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
Time Frame: Week 5 of each treatment period
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Amantadine | Modafinil | Methylphenidate
Number analyzed (Participants) | 123 | 124 | 124 | 127
score on a scale | 9.4 [8.7 to 10.1] | 9.3 [8.6 to 10.1] | 8.3 [7.6 to 9.1] | 8.8 [8.1 to 9.6]

4. Post Hoc Outcome: Acceptability of Treatment as Assessed by a Single Question Questionnaire
Description: Participants will answer yes or no to this question: "Taken into consideration the possible benefits and/or disadvantages of this medication, would you choose it, going forward to treat your MS fatigue?". The number of participants who answered "Yes" to this question is reported here.
Time Frame: Week 5 of each treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Amantadine | Modafinil | Methylphenidate
Number analyzed (Participants) | 123 | 124 | 124 | 127
Participants | 39 | 41 | 55 | 55

ADVERSE EVENTS:
Time Frame: Adverse events were collected during each six-week medication period.
Description: The numbers in the adverse event section are patients who constitute the safety dataset. These are patients who at least took one dose of that medication (whether or not they had their efficacy measured).
Arm/Group | Placebo | Amantadine | Modafinil | Methylphenidate
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/127 | 0/125 | 0/129
Serious Adverse Events (participants affected / at risk) | 0/124 | 2/127 | 1/125 | 0/129
Other Adverse Events (participants affected / at risk) | 38/124 | 49/127 | 50/125 | 51/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=124) | Amantadine (N=127) | Modafinil (N=125) | Methylphenidate (N=129)
Pulmonary embolism (Vascular disorders) | 0 | 1 | 0 | 0
Myocardiitis (Cardiac disorders) | 0 | 1 | 0 | 0
MS exacerbation (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=124) | Amantadine (N=127) | Modafinil (N=125) | Methylphenidate (N=129)
Cardiac disorders (Cardiac disorders) | 3 | 3 | 2 | 4
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Eye disorders (Eye disorders) | 0 | 1 | 2 | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 10 | 14 | 19 | 13
General disorders (General disorders) | 2 | 4 | 5 | 4
Immune system disorders (Immune system disorders) | 0 | 1 | 1 | 0
Infections and infestations (Infections and infestations) | 3 | 2 | 2 | 1
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 4
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 | 1 | 3 | 0
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 1
Nervous system disorders (Nervous system disorders) | 13 | 24 | 22 | 20
Psychiatric disorders (Psychiatric disorders) | 10 | 20 | 18 | 23
Renal and urinary disorders (Renal and urinary disorders) | 0 | 0 | 1 | 0
Reproductive system (Reproductive system and breast disorders) | 1 | 1 | 2 | 2
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 2
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 | 2 | 5 | 0
Vascular disorders (Vascular disorders) | 1 | 3 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT03185065/Prot_SAP_000.pdf